CLINICAL TRIAL: NCT02577120
Title: Wound Healing Endpoint and Recurrence
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sashwati Roy (Other)
Responsible Party: Sponsor-Investigator, Sashwati Roy, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY24010050
Record Dates: First submitted 2015-06-26; First posted 2015-10-16 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Wound; Burn Wound; Diabetic Foot Ulcers; Pressure Ulcers; Venous Leg Ulcers; Chronic; Wound
Keywords: Epiceram
MeSH Terms: conditions — Burns; Diabetic Foot; Pressure Ulcer; Bronchiolitis Obliterans Syndrome; Wounds and Injuries | interventions — Petroleum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TEWL - Epiceram (Experimental): Subjects will have the TEWL reading completed at the wound site and a control site (anatomically matched site on the patients contralateral side) at the second study visit. If the wound site reading is less than 3 times the value of the control site subjects
  Interventions: Device: Epiceram Skin Barrier Function
- TEWL - Vaseline Petroleum Jelly (Placebo Comparator): Subjects will have the TEWL reading completed at the wound site and a control site (anatomically matched site on the patients contralateral side) at the second study visit. If the wound site reading is less than 3 times the value of the control site subjects
  Interventions: Biological: Vaseline Petroleum Jelly

INTERVENTIONS:
Device: Epiceram Skin Barrier Function — Epiceram is a non-sterile, viscous, lipid-rich emulsion
  Other Names: Epiceram
  Arms: TEWL - Epiceram
Biological: Vaseline Petroleum Jelly — A skin protectant used for temporarily protecting minor cuts, scraps, burns, and helps to protect and help relieve chapped or cracked skin and lips.
  Other Names: Petroleum
  Arms: TEWL - Vaseline Petroleum Jelly

SUMMARY:
This study is a continuation of a previously approved protocol conducted at Ohio State University and Indiana University. The first two aims of the original protocol have been completed, and this protocol will finish enrollment for the third aim, comparing Hi TEWL and Low TEWL measurements, and whether a HiTEWLmeasurement indicates a seemingly healed wound is more likely to recur/reopen toa new wound.

Of the 105 desired subjects, 62 subjects have already been recruited and completed their study participation at the previous university. 43 additional subjects will be recruited to complete the enrollment goal here at the University of Pittsburgh.

DETAILED DESCRIPTION:
In the United States, chronic wounds represent a major public health burden. Estimates put the number of chronic wounds cases at over 6.5 million with a cost burden of over $50 billion14. According to the current standard of care (SoC), wound closure is assessed visually. The FDA defines complete wound closure of chronic non-healing wounds as "skin closure (as assessed visually) without drainage or dressing requirements identified at two consecutive study visits that are 2 weeks apart" and requires therapeutic trials for chronic wounds to be designed such that the enrolled patients will be evaluated for at least 3 months following completeclosure19.

The expectation is that successful intervention should keep the wound closed for at least 90 days. This study contends that visual inspection of wounds is insufficient to certify closure - a critical endpoint that drives treatment decisions. Considering that almost two-thirds of all chronic wounds are estimated to be biofilminfected6, and the observation that biofilm-infected wounds may be visually closed but functionally (barrier function) open, the significance of the proposed hypothesis is substantial.

The proposed study has the clear potential to lay a strong rationale that would potentially change the wound care paradigm by requiring that measurement of skin barrier function be the new endpoint to define wound closure. Reported recurrence rates for most chronic ulcer types remain extremely high, ranging from 40-79%4,5, 24%-57% for venous ulcers, and upward of 60% for diabetic ulcers supporting the importance of preventive efforts1,2. In that context it is of extraordinary significance to ask whether "defective closure" (visually closed with TEWL (Trans-Epidermal Water Loss) >3x the value of intact skin; high TEWL) predicts poor post-closure outcome e.g. recurrence. These questions may only be meaningfully asked in a patient-based pilot and that is exactly the intent of Aim 2. Findings of the proposed pilot will inform a larger future trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Willing to comply with protocol instructions, including all study visits and study activities.
3. One of the following: Healed wound (within 10 days prior to consent/screening visit) that was previously a chronic wound of multiple etiologies and open for at least30 days, including:

   i. Diabetic foot ulcers, Wagner grade 1-3 ii. Pressure ulcers, stage 2-3 iii. Venous leg ulcers, confirmed by venous duplex iv. Burn wounds
4. If candidate has a diabetic foot ulcer, ABI score measurement at Visit 1 must be between 0.7 and 1.2. If score is below or above, candidate will be considered a screen fail. Score can be gathered from EMR in previous 3 months to visit 1 if done as SOC or completed during visit 1.

Exclusion Criteria:

1. Individuals who are deemed unable to understand the procedures, risks and benefits of the study, (i.e. unable to provide informed consent).
2. Subjects with marked immunodeficiency (HIV/AIDS, organ transplant patients and cancer patients and patients with autoimmune disease on immunosuppressive medications).
3. Wounds closed or to be closed by flap or graft coverage - including stage 4pressure ulcers and Wagner grade 4 or 5 diabetic foot ulcers.
4. Prisoners
5. Patients with allergies to petrolatum
6. Patients who are currently enrolled in another research study which includes investigational treatment and/or medication
7. Patients with an HbA1c score greater than 10.0 at Visit 1, will be considered a screen fail. Score can be gathered from EMR in previous 12 months to visit 1 if done as SOC, or completed during visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
TEWL | 12 weeks
  If topical application of the FDA approved EpiCeram® restores barrier function (TEWL) defectively closed wounds. These will be compared to a Placebo cream, Vaseline and will be seen after 3 months of application to the wound site.

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Pittsburgh / McKeesport Clinic, Pittsburgh, Pennsylvania
  - University of Pittsburgh / Mercy Clinic, Pittsburgh, Pennsylvania
  - University of Pittsburgh / Passavant, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Final processed data will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 8, 2019 - December 31, 2027
Access Criteria: Data will be made available by the PI per Institution sharing policy and via published paper.
URL: https://www.ncbi.nlm.nih.gov/pmc/about/public-access-info/

REFERENCES:
- [Background] Apelqvist J, Larsson J, Agardh CD. Long-term prognosis for diabetic patients with foot ulcers. J Intern Med. 1993 Jun;233(6):485-91. doi: 10.1111/j.1365-2796.1993.tb01003.x. PMID 8501419
- [Background] Barwell JR, Taylor M, Deacon J, Ghauri AS, Wakely C, Phillips LK, Whyman MR, Poskitt KR. Surgical correction of isolated superficial venous reflux reduces long-term recurrence rate in chronic venous leg ulcers. Eur J Vasc Endovasc Surg. 2000 Oct;20(4):363-8. doi: 10.1053/ejvs.2000.1196. PMID 11035968
- [Background] Brooks B, Dean R, Patel S, Wu B, Molyneaux L, Yue DK. TBI or not TBI: that is the question. Is it better to measure toe pressure than ankle pressure in diabetic patients? Diabet Med. 2001 Jul;18(7):528-32. doi: 10.1046/j.1464-5491.2001.00493.x. PMID 11553180
- [Background] Chamlin SL, Kao J, Frieden IJ, Sheu MY, Fowler AJ, Fluhr JW, Williams ML, Elias PM. Ceramide-dominant barrier repair lipids alleviate childhood atopic dermatitis: changes in barrier function provide a sensitive indicator of disease activity. J Am Acad Dermatol. 2002 Aug;47(2):198-208. doi: 10.1067/mjd.2002.124617. PMID 12140465
- [Background] Disa JJ, Carlton JM, Goldberg NH. Efficacy of operative cure in pressure sore patients. Plast Reconstr Surg. 1992 Feb;89(2):272-8. doi: 10.1097/00006534-199202000-00012. PMID 1732895
- [Background] Goodman CM, Cohen V, Armenta A, Thornby J, Netscher DT. Evaluation of results and treatment variables for pressure ulcers in 48 veteran spinal cord-injured patients. Ann Plast Surg. 1999 Jun;42(6):665-72. doi: 10.1097/00000637-199906000-00015. PMID 10382806
- [Background] James GA, Swogger E, Wolcott R, Pulcini Ed, Secor P, Sestrich J, Costerton JW, Stewart PS. Biofilms in chronic wounds. Wound Repair Regen. 2008 Jan-Feb;16(1):37-44. doi: 10.1111/j.1524-475X.2007.00321.x. Epub 2007 Dec 13. PMID 18086294
- [Background] Lavrijsen AP, Higounenc IM, Weerheim A, Oestmann E, Tuinenburg EE, Bodde HE, Ponec M. Validation of an in vivo extraction method for human stratum corneum ceramides. Arch Dermatol Res. 1994;286(8):495-503. doi: 10.1007/BF00371579. PMID 7864665
- [Background] Lopez D, Vlamakis H, Kolter R. Generation of multiple cell types in Bacillus subtilis. FEMS Microbiol Rev. 2009 Jan;33(1):152-63. doi: 10.1111/j.1574-6976.2008.00148.x. Epub 2008 Nov 19. PMID 19054118
- [Background] Park SC, Choi CY, Ha YI, Yang HE. Utility of Toe-brachial Index for Diagnosis of Peripheral Artery Disease. Arch Plast Surg. 2012 May;39(3):227-31. doi: 10.5999/aps.2012.39.3.227. Epub 2012 May 10. PMID 22783531
- [Background] Pinnagoda J, Tupker RA, Agner T, Serup J. Guidelines for transepidermal water loss (TEWL) measurement. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1990 Mar;22(3):164-78. doi: 10.1111/j.1600-0536.1990.tb01553.x. PMID 2335090
- [Background] Romanos MT, Raspovic A, Perrin BM. The reliability of toe systolic pressure and the toe brachial index in patients with diabetes. J Foot Ankle Res. 2010 Dec 22;3:31. doi: 10.1186/1757-1146-3-31. PMID 21176166
- [Background] Roy S, Elgharably H, Sinha M, Ganesh K, Chaney S, Mann E, Miller C, Khanna S, Bergdall VK, Powell HM, Cook CH, Gordillo GM, Wozniak DJ, Sen CK. Mixed-species biofilm compromises wound healing by disrupting epidermal barrier function. J Pathol. 2014 Aug;233(4):331-343. doi: 10.1002/path.4360. Epub 2014 May 27. PMID 24771509
- [Background] Roy S, Patel D, Khanna S, Gordillo GM, Biswas S, Friedman A, Sen CK. Transcriptome-wide analysis of blood vessels laser captured from human skin and chronic wound-edge tissue. Proc Natl Acad Sci U S A. 2007 Sep 4;104(36):14472-7. doi: 10.1073/pnas.0706793104. Epub 2007 Aug 29. PMID 17728400
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] Smack DP, Harrington AC, Dunn C, Howard RS, Szkutnik AJ, Krivda SJ, Caldwell JB, James WD. Infection and allergy incidence in ambulatory surgery patients using white petrolatum vs bacitracin ointment. A randomized controlled trial. JAMA. 1996 Sep 25;276(12):972-7. PMID 8805732
- [Background] Tetteh HA, Groth SS, Kast T, Whitson BA, Radosevich DM, Klopp AC, D'Cunha J, Maddaus MA, Andrade RS. Primary palmoplantar hyperhidrosis and thoracoscopic sympathectomy: a new objective assessment method. Ann Thorac Surg. 2009 Jan;87(1):267-74; discussion 274-5. doi: 10.1016/j.athoracsur.2008.10.028. PMID 19101310
- [Background] Thiele JJ, Traber MG, Packer L. Depletion of human stratum corneum vitamin E: an early and sensitive in vivo marker of UV induced photo-oxidation. J Invest Dermatol. 1998 May;110(5):756-61. doi: 10.1046/j.1523-1747.1998.00169.x. PMID 9579541
- [Background] Thiele JJ, Traber MG, Polefka TG, Cross CE, Packer L. Ozone-exposure depletes vitamin E and induces lipid peroxidation in murine stratum corneum. J Invest Dermatol. 1997 May;108(5):753-7. doi: 10.1111/1523-1747.ep12292144. PMID 9129228
- [Background] FDA Wound Healing Clinical Focus Group.. Guidance for industry: chronic cutaneous ulcer and burn wounds-developing products for treatment. Wound Repair Regen. 2001 Jul-Aug;9(4):258-68. doi: 10.1046/j.1524-475x.2001.00258.x. No abstract available. PMID 11679134
- [Derived] Sen CK, Roy S, Mathew-Steiner SS, Gordillo GM. Biofilm Management in Wound Care. Plast Reconstr Surg. 2021 Aug 1;148(2):275e-288e. doi: 10.1097/PRS.0000000000008142. PMID 34398099